CLINICAL TRIAL: NCT03529175
Title: Randomised Phase II Trial to Investigate Two Different Schedules of Nab-paclitaxel (Abraxane) Combined With Gemcitabine as First Line Treatment for Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Scheduling Nab-paclitaxel With Gemcitabine
Acronym: SIEGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, CCTU-Cancer Theme, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIEGE (AX-PANC-PI-0101)
Record Dates: First submitted 2014-05-01; First posted 2018-05-18 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Pancreatic Adenocarcinoma Metastatic
MeSH Terms: interventions — Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concomitant (Active Comparator): Intravenous Abraxane125 mg/m2 30-minute infusion followed immediately by intravenous Gemcitabine 1000 mg/m2 30-minute infusion will be administered on days 1, 8 and 15 of a 4-week cycle.
  Interventions: Drug: Abraxane (nab-paclitaxel); Drug: Gemcitabine
- Sequential (Active Comparator): Intravenous Abraxane 125 mg/m2 30-minute infusion will be administered on days 1, 8 and 15 of a 4-week cycle. Intravenous Gemcitabine 1000 mg/m2 30-minute infusion will be administered on days 2, 9 and 16 of a 4-week cycle. Gemcitabine must be delivered 24 +/- 2 hours after commencing Abraxane infusion.
  Interventions: Drug: Abraxane (nab-paclitaxel); Drug: Gemcitabine

INTERVENTIONS:
Drug: Abraxane (nab-paclitaxel)
Drug: Gemcitabine

SUMMARY:
Metastatic pancreatic cancer is difficult to treat. Until recently, most patients would be offered treatment with a chemotherapy drug called gemcitabine. However, a large international trial showed that combining gemcitabine with a drug called nab-paclitaxel (or abraxane) was more effective compared with gemcitabine alone. The purpose of this study is to compare two different ways of combining gemcitabine with abraxane. Conventionally, both drugs are given on the same day via a drip into a vein in the arm but research suggests that giving abraxane 24 hours in advance of gemcitabine could possibly be more beneficial.

In this study, blood and tumour samples will be collected and analysed to try to confirm what has been seen in the laboratory studies. In addition, the investigators wish to find out whether certain tumour characteristics (called biomarkers) can be used to predict for response to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Signed informed consent and ability to comply with the protocol
* Histologically or cytologically confirmed metastatic PDAC
* Radiologically confirmed stage IV disease and measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1; baseline tumour assessments and measurements must be done within 28 days prior to randomisation
* Karnofsky performance status ≥70%
* Life expectancy >12 weeks from the date of screening assessment
* Adequate bone marrow function

  * Absolute neutrophil count (ANC) ≥1.5 x 109 /L
  * Haemoglobin (Hb) ≥ 100 g/L
  * Platelets ≥100 x 109 /L
  * White blood cell count (WBC) ≥ 3 x 109 /L
* Adequate liver function

  * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤2.5 x upper limit of normal range (ULN)
  * Total bilirubin <1.5 x ULN
* Adequate renal function defined as a serum creatinine ≤1.5 x ULN or calculated creatinine clearance by Cockcroft-Gault of ≥50 mL/min
* Received no prior systemic therapy for metastatic disease
* Prior adjuvant chemotherapy (with GEM or any other drug/s) is allowed if completed at least 6 months previously
* Prior radiotherapy is allowed as long as there is measurable disease which has not been irradiated
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, completion of QoL and HE questionnaires and other study procedures
* Confirmation of tumour tissue sample collected within 12 weeks prior to randomisation and blood to be taken prior to randomisation
* Women of child-bearing potential (WCBP), defined as a sexually mature woman not surgically sterilized or not post-menopausal for at least 24 consecutive months if age ≤55 years or 12 months if age >55 years, must have a negative serum or urine pregnancy test within 14 days prior to randomisation
* All WCBP and all sexually active male patients must agree to use effective contraception methods throughout the study and for 30 days after the final dose of study drug for WCBP and for up to 6 months after treatment for male patients

Exclusion Criteria:

* Patients with operable or locally advanced PDAC
* Other invasive malignancies diagnosed within the last 5 years, except non-melanoma skin cancer and localized cured prostate cancer
* Significant acute or chronic medical or psychiatric condition, disease or laboratory abnormality which in the judgment of the investigator would place the patient at undue risk or interfere with the trial. Examples include, but are not limited to:

  * Patients who have had a venous thromboembolic event who are not appropriately anticoagulated or have had a significant bleeding episode in the 3 weeks prior to randomisation
  * Patients with symptoms of severe chronic obstructive airways disease or significant shortness of breath at rest AND have an FEV1<1.0 L within the last 6 months
  * Patients with a history of interstitial lung disease, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis, cystic fibrosis or bronchiectasis
  * Patients with uncontrolled ischaemic heart or other cardiovascular event (myocardial infarction (MI), new angina, stroke transient ischaemic attack (TIA), or new congestive cardiac failure (CCF)) within the last 6 months
  * Patients with stable but significant cardiovascular disease defined by heart failure (New York Heart Association Functional Classification (NYHF) III or IV, see Appendix 3) or frequent angina
  * Presence of active infection
  * Cirrhotic liver disease, known chronic active or acute hepatitis B, or hepatitis C
  * Known allergy or hypersensitivity to GEM or ABX
* Women who are pregnant, plan to become pregnant or are lactating
* Routine use of any of the following will exclude patients:

  * Oral anti-oxidant supplements: beta-carotene, selenium, lutein, zeaxanthin, lycopene, pycnogenol, fernblock, omega-3S, vitamin C, vitamin E, astaxanthin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival | From participant randomisation to the point at which disease progression is reported (i.e. 12 months)
  The primary objective of the trial is to investigate the outcome of sequential administration of nab-paclitaxel combined with gemcitabine (ABX/GEM, 24 hours apart) in patients with metastatic pancreatic ductal adenocarcinoma (PDAC) in terms of progression-free survival.

SECONDARY OUTCOMES:
Patient Safety | 1 year after end of treatment visit
  Adverse Events (including Serious Adverse Events), abnormal laboratory test results and performance status
Treatment Efficacy | 8 weeks
  response to treatment assessed using radiological RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Pippa Corrie, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital
Locations (23):
- United Kingdom (23):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - Peterborough City Hospital, Peterborough, Cambridgeshire
  - Ysbyty Gwynedd, Bangor
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Haematology & Oncology Centre, Bristol
  - Velindre Cancer Centre, Cardiff
  - Colchester Hospital, Colchester
  - University Hospitals Coventry & Warwickshire, Coventry
  - Edinburgh Cancer Research Centre, Edinburgh
  - The Beatson Oncology Centre, Glasgow
  - The Royal Surrey County Hospital, Guildford
  - St James' Institute of Oncology, Leeds
  - Leicester Royal Infirmary, Leicester
  - Clatterbridge Cancer Centre, Liverpool
  - Barts Health NHS Trust, London
  - Hammersmith Hospital, London
  - The Royal Free Hospital, London
  - University College London Hospital, London
  - The Christie Hospital, Manchester
  - Churchill Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Dayimu A, Di Lisio L, Anand S, Roca-Carreras I, Qian W, Al-Mohammad A, Basu B, Valle JW, Jodrell D, Demiris N, Corrie P. Clinical and biological markers predictive of treatment response associated with metastatic pancreatic adenocarcinoma. Br J Cancer. 2023 May;128(9):1672-1680. doi: 10.1038/s41416-023-02170-9. Epub 2023 Feb 22. PMID 36813867
- [Derived] Corrie PG, Qian W, Basu B, Valle JW, Falk S, Lwuji C, Wasan H, Palmer D, Scott-Brown M, Wadsley J, Arif S, Bridgewater J, Propper D, Gillmore R, Gopinathan A, Skells R, Bundi P, Brais R, Dalchau K, Bax L, Chhabra A, Machin A, Dayim A, McAdam K, Cummins S, Wall L, Ellis R, Anthoney A, Evans J, Ma YT, Isherwood C, Neesse A, Tuveson D, Jodrell DI. Scheduling nab-paclitaxel combined with gemcitabine as first-line treatment for metastatic pancreatic adenocarcinoma. Br J Cancer. 2020 Jun;122(12):1760-1768. doi: 10.1038/s41416-020-0846-2. Epub 2020 Apr 30. PMID 32350413
- See also: University of Cambridge Pancreatic Cancer Centre — http://www.cambridge-pcc.org/trials.html